CLINICAL TRIAL: NCT06113497
Title: A Prospective Study on the Comparison of Postoperative Pain According to the Use of Cocktail Therapy in Laminoplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Kyung-Chung Kang, Associate Professor, Spine Center, Department of Orthopaedic Surgery, Kyunghee University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: futurespine
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Adverse Effects in the Therapeutic Use of Analgesic, Antipyretic and Anti-Inflammatory Drug, Unspecified
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): The group that received normal saline 40ml injection into the deep fascia and muscular layer during wound closure.
- Group 2 (Experimental): The group that received cocktail therapy injection into the deep fascia and muscular layer during wound closure.
  Interventions: Drug: Cocktail injection

INTERVENTIONS:
Drug: Cocktail injection — Morphine 5 mg, ropivacaine 150 mg, tramadol 40 mg, epinephrine 1 mg, ketorolac 60 mg, and ketamine 1 g will be mixed with normal saline to prepare a total volume of 60 ml
  Other Names: Normal saline injection
  Arms: Group 2

SUMMARY:
This study is the first prospective randomized controlled trial to analyze the effects and safety of multimodal cocktail injections after cervical laminoplasty

DETAILED DESCRIPTION:
This study is the first prospective randomized controlled trial to analyze the effects and safety of multimodal cocktail injections after cervical laminoplasty. Through this study, we anticipate that the potential usefulness of multimodal cocktail analgesic injections in various aspects of spinal surgery will be demonstrated, offering valuable insights and possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical myelopathy or radiculopathy and scheduled to undergo laminoplasty
* Recorded preoperative upper limb pain (Visual Analog Scale [- VAS] ), neck pain (VAS), Japanese Orthopaedic Association (JOA) scores, and Neck Disability Index (NDI) scores.
* Adults aged 20 years and above, but below 80 years capable of articulating their own pain or functional abnormalities
* Cognitive function at a level that enables them to comprehend and adhere to study procedures

Exclusion Criteria:

* Previous surgical treatment of the cervical spine.
* Adolescents aged 20 years or below, pregnant individuals, or those with the potential for pregnancy.
* Hypersensitivity reactions to mixed medications used in Cocktail therapy. (morphine 5 mg, ropiva 150 mg, tamceton 40 mg, epinephrine 1 mg, ketocin 60 mg, jetiam 1 g).
* Patients who lack the capacity for medical consent or are unable to communicate effectively in a medical context.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-10-24 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain (VAS/Visual Analog Score) | Baseline and Post operation 7 days
  A VAS score, also known as a Visual Analog Scale score, is a common method used in healthcare and research to measure subjective or self-reported sensations or experiences, such as pain, anxiety, mood, or other subjective states. It typically consists of a horizontal or vertical line, usually 10 centimeters in length, with anchor points at either end. One end is labeled with the most negative or extreme aspect of the sensation or experience being measured, and the other end is labeled with the most positive or least extreme aspect.
Change from Baseline in function (JOA/Japanese Orthopaedic Association Score) score | Baseline and Post operation 7 days
  The JOA score is often calculated based on a specific set of criteria and is used to help guide treatment decisions and monitor a patient's progress. It provides a standardized way to assess and communicate the clinical status of individuals with cervical myelopathy. The score may range from 0 (severe impairment) to 17 (normal function), with lower scores indicating greater disability.
Change from Baseline in function (NDI/Neck Disability Index score) score | Baseline and Post operation 7 days
  The NDI questionnaire typically consists of ten questions or items, and individuals are asked to rate their level of disability or limitation in various aspects of daily life due to neck pain. The questions cover a range of activities, including personal care, work, sleep, and recreational activities. Each question is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating severe disability. The individual's responses to these questions are then totaled to calculate the NDI score, usually expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Chung Kang, Associate Professor, Study Chair — Kyunghee University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soh J, Park HS, Lee WY, Park SH, Kang KC. The effects of multimodal cocktail analgesic local injection in postoperative pain control after laminoplasty: A study protocol of a prospective randomized controlled trial. PLoS One. 2025 Jun 13;20(6):e0324791. doi: 10.1371/journal.pone.0324791. eCollection 2025. PMID 40512737